CLINICAL TRIAL: NCT06684782
Title: Prevalence and Characteristics of Restless Leg Syndrome in Thai Patients With Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Jindapa Srikajon, MD., Siriraj Hospital
Other Study IDs: 762/2567(IRB1)
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Restless Legs Syndrome
Keywords: restless leg syndrome; parkinson's disease; prevalence; Thai population
MeSH Terms: conditions — Restless Legs Syndrome; Parkinson Disease | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with parkinson's disease
  Interventions: Other: Screening for symptoms of restless leg syndrome

INTERVENTIONS:
Other: Screening for symptoms of restless leg syndrome — The patients will be screened for restless leg syndrome by clinical questioning.

SUMMARY:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by pathologic intraneuronal alpha-synuclein-positive Lewy bodies and neuronal cell loss. The cardinal clinical symptoms and signs of PD are bradykinesia, rigidity, tremor, postural instability, and freezing attacks. The prevalence of PD increases with age, affecting 1-2% of the population over the age of 65 years, and 3% of those over 85 years.

Restless legs syndrome (RLS) represents disturbing symptoms in lower limbs that lead to the urge to move, occurring in rest periods. Movements can partially or completely relieve these abnormal feelings. In 2014, the International RLS Study Group (IRLSSG) established five mandatory criteria for the diagnosis of RLS. Several studies supported that RLS and PD may share pathophysiological mechanisms.

DETAILED DESCRIPTION:
In the general population, the prevalence of RLS was reported to be up to 10%. In Parkinson's disease (PD), the mean prevalence of RLS was 15.74%. Cross-sectional studies show a variable prevalence of RLS in PD patients ranging approximately from 0 to 50%. In case-control studies, the mean prevalence of RLS was higher in people with PD (12%) vs. healthy controls (5.1%). One four-year longitudinal study reported an increase in RLS prevalence from 4.6% to 16.3% along with disease progression. Interestingly, RLS was found to have various prevalence depending on geographic areas: highest in European populations (5% to 12%), intermediate in Asian countries (1% to 8%), and lowest in African countries (<1%).

In Patients with Parkinson's disease, diagnosis of RLS is challenging due to multiple confounders such as motor fluctuations, akathisia, etc. It is crucial to pick up RLS in Parkinson's disease and properly manage the symptoms. RLS not only causes impaired quality of life but also possibly leads to cardiovascular consequences. RLS was associated with statistically significantly less future cardiovascular risk in RLS patients with treatment than in those without treatment. Nevertheless, there have been no consistent studies of this association in Parkinson's disease yet.

From the literature review, very few data have been stated regarding RLS in Thai patients with Parkinson's disease. There was only one study focusing on the prevalence of RLS in Thailand, in which the prevalence of RLS in Thai Parkinson's patients was only 1.6%. According to the author, there were possible explanations for the low prevalence. Firstly, they only included participants with idiopathic RLS. Secondly, high doses of dopaminergic agents might obscure the symptoms of RLS in those patients with Parkinson's disease. Moreover, they screened patients with the Cambridge-Hopkins diagnostic questionnaire which had not been validated in Thai people yet. For all these reasons, we believe that the prevalence of RLS in Thai patients with Parkinson's disease would be different with another methodology. We also would like to know more about the characteristics of RLS in Thai Parkinson's disease patients, which might help improve RLS detection in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease aged from 18 to 80 years who met the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Diagnostic criteria.

Exclusion Criteria:

* Patients with atypical or secondary parkinsonism.
* Patients with Mini-mental status exam (MMSE) less than 24 of 30.
* Patients with secondary causes of restless leg syndrome including end-stage renal disease, iron deficiency anemia and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease aged from 18 to 80 years who met the UK Parkinson's Disease Society Brain Bank Diagnostic Criteria. The patients must regularly visit the movement disorders clinic at least 2 times per year.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence of restless leg syndrome in patients with Parkinson's disease | At the time of recruitment

SECONDARY OUTCOMES:
Clinical characteristics of Parkinson's disease patients with restless leg syndrome | At the time of recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Jindapa Srikajon, Doctor of Medicine, Principal Investigator — Siriraj Sleep Center, Faculty of Medicine, Siriraj Hospital, Mahidol University
Locations (2):
- Thailand (2):
  - Siriraj Hospital, Mahidol University, Bangkok, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided